CLINICAL TRIAL: NCT07062575
Title: Clinical Investigation on the Safety and Performance of the ABLE Daily to Assist People With Spinal Cord Injury in Performing Ambulatory Functions in Home and Community Settings
Brief Title: Exoskeleton Training at Home to Assist Participants With Spinal Cord Injuries to Perform Ambulatory Functions.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was temporarily halted on January 13th, 2026, to investigate a technical device performance issue. This preventive action is not related to safety concerns, and no increased risk to participants has been identified.
Sponsor: ABLE Human Motion S.L. (Industry)
Collaborators: Sint Maartenskliniek (Other); Universitat Politècnica de Catalunya (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ABLEdailySCI; CIV-25-01-050614 (Other: CCMO)
Record Dates: First submitted 2025-05-26; First posted 2025-07-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with exoskeleton (Experimental): The participants will receive training sessions with the ABLE Daily at Sint Maartenskliniek. After they pass the skills and knowledge exam, they will receive the ABLE Daily at their disposal at home for twelve weeks.
  Interventions: Device: ABLE Daily

INTERVENTIONS:
Device: ABLE Daily — The participants will receive training sessions with the ABLE Daily at Sint Maartenskliniek. After they pass the skills and knowledge exam, they will receive the ABLE Daily at their disposal at home for twelve weeks

SUMMARY:
The goal of this clinical trial is to to confirm the safety and performance of the ABLE Daily to perform ambulatory functions in home and community settings for people with spinal cord injury.

The experimental period will cover the training period with the ABLE Daily exoskeleton (3 weeks of use at the investigational site with a total of 9 sessions) and the home period (12 weeks of personal use at home and community environments).

DETAILED DESCRIPTION:
The ABLE Daily Exoskeleton is a wearable powered lower-limb exoskeleton that actively assists individuals with spinal cord injury to stand up, walk, ascend and descend a ramp of 5 degrees and sit down. The device consists of a rigid brace that attaches to the torso, legs and feet of the user via straps and supports. It is a bilateral robotic exoskeleton with four battery-powered motors that drive the knee and hip joints assisting in flexion-extension. The other degrees of freedom of the hip and knee joints are restricted. The ankle joint of the exoskeleton is passively articulated with a spring within a limited range of motion.

The experimental period will cover the training period happening at the investigational site where the participants and their companions will be trained 3 times a week. They will then have to perform a community skills test, if passed they will be allowed to take the exoskeleton home and use it in their daily life for 12 weeks. Pre and post assessments will be made.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Chronic SCI (>6 months)
* Injury at levels T1 to L5 (AIS A to D)
* Walking Index for Spinal Cord Injury (WISCI) score 0 until 9
* Height between 150-200 cm
* Weight less than 100 kg
* Capable of giving informed consent on their own
* Able to train (at least) 3 days/week
* Able to have at least 1 companion / buddy who can attend a minimum of two of the training sessions, besides the final assessment, and who will learn how to assist them at home and in the community (ideally two companions)
* Proficiency in walking with the ABLE Exoskeleton
* At least 8 weeks with minimal use (less than 5 sessions) of wearable robotic exoskeletons for gait assistance at the start of the study.

Exclusion Criteria:

* High risk of fractures due to osteoporosis, a dual energy X-ray absorptiometry (DEXA)-scan at the hip, distal femur, and proximal tibia BMD score
* Fragility fractures of the lower limbs in the last 2 years
* Deterioration >3 in the International Standards for Neurological Classification of SCI (ISNCSCI) score in the last 4 weeks
* Spinal instability, like spondylolisthesis
* Disorders of the arms and hands that make walking with crutches impossible
* Modified Ashworth Scale (MAS) >3 in lower limbs
* Cardiovascular health issues which prevent the participant from training
* Instability to tolerate 10 minutes of standing without clinical symptoms of orthostatic hypotension
* Psychological, cognitive issues, or any other condition that does not allow a participant to follow study procedures
* Medically unstable due to severe comorbidities, including any condition that a physician deems inappropriate for completing study participation
* Skin problems in areas that would be in contact with the device
* Height, width, weight, or other anatomical limitations (such as differences in leg length) incompatible with the device
* Insufficient joint range of motion (ROM) for the device
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of the device | Through study completion (up to 16 weeks)
  The total number of adverse events and serious adverse events related to the investigational device at the end of the study will be measured.
Performance of the device during the training period | Through the training period (up to 3 weeks) from training session 1-9
  The number and type of device errors or use errors during the training period.
Performance of the device in the home/community period | Through the home/community period (up to 12 weeks)
  The amount of use of the device during the home/community use period, as measured by the number of sessions and the walking time, number of steps, and distance walked per session.
Performance of the device in the home/community period | Through the home/community period (up to 12 weeks)
  The usability of the device as measured by the purpose and location of use of the device during the home/community use period which will be registered in a logbook by the participant.
Performance of the device in the home/community period | Through the home/community period (up to 12 weeks)
  The number and type of device errors at the end of the home/community use period will be registered.

SECONDARY OUTCOMES:
Perceived health status | At baseline and the final assessment at end of the study (16 weeks)
  The change from baseline to final assessment of the overall perceived health status of the participants, as measured by the scores of the 36-Item Short Form Survey Instrument (SF-36).
  Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to high Quality of Life. Lower scores indicate more disability, while higher scores indicate less disability.
Gait performance while using the device (6MWT) | After training period (3 weeks) and at the final assessment at the end of the study (16 weeks)
  The change from the Community Skills Test to the final exoskeleton assessment of the 6-Minute Walk Test (6MWT). The outcome will be the distance walked during the 6 minutes after the training period and once again after the home period.
User satisfaction | At the final assessment at the end of the study (16 weeks)
  The general user satisfaction of participants, companions, and therapists at the end of the study, as measured by the scores of the Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0).
  12 item instrument used to assess satisfaction with a specific assistive device; eight of these items assess characteristics of that assistive device and the remaining four items assess service and include:
  1. Service delivery
  2. Repairs and service of the device
  3. Professionalism of service
  4. Follow-up service Participants are asked to rate their satisfaction for the device on a five point scale that ranges from "not satisfied" at all to "very satisfied." Finally, participants are asked to choose the three most important items related to the assistive device in question System Usability Scale (SUS) to measure the perceived usability of the device. The scales value from 0 to 4 (with four being the most positive response).
Gait performance using the device: 10-Meter Walk Test (10MWT) | After training period (3 weeks) and at the final assessment at the end of the study (16 weeks)
  The 10 meter walk test will be used to compare performance after the training period and once again after the home period to monitor any changes in speed.

OTHER OUTCOMES:
Cardiovascular health | Baseline assessment and at the final assessment at the end of the study (16 weeks)
  Blood draw test to check levels of high-density lipoprotein cholesterol (HDL-c), Low-Density Lipoprotein Cholesterol (LDL-c), Triglyceride (TG), and Total Cholesterol (TC).
  Improvement is indicated with lower values of LDL-c and lower Triglycerides
Respiratory Parameters | Baseline assessment, during the 6 minute walk test and at the final assessment at the end of the study (16 weeks)
  Spirometry to assess the force vital capacity (FVC). FVC is crucial for evaluating lung function and respiratory and global health. Improvement indicates higher values of FVC.
Spasticity | Baseline assessment, end of training period (3 weeks), final assessment at the end of the study (16 weeks)
  Visual analog scale (VAS) is a self-report tool that allows individuals to rate their perceived level of spasticity on a continuous scale, typically ranging from 0 to 10, where higher scores indicate greater severity. Spasticity is a complex phenomenon that can vary greatly in intensity and impact from person to person. The VAS provides a means for individuals to subjectively quantify and communicate their experience of spasticity, capturing nuances that may not be fully captured by objective measures alone. 0 indicated no spasticity and 10 indicates the most spasticity experienced.
Bowel and bladder management (SCI-QOL) | Baseline assessment and at the final assessment at the end of the study (16 weeks)
  Bladder Management Difficulties and Bowel Management Difficulties items from the Spinal Cord Injury - Quality of Life (SCI-QOL) questionnaire. The SCI-QOL questionnaire is a validated measure specifically designed to assess the quality of life in individuals with SCI across various domains, including bladder and bowel function
Body composition using BMI | Baseline assessment and at the final assessment at the end of the study (16 weeks)
  Body weight provides valuable information about body composition.
  Body Mass Index (BMI) is a simple and straightforward measure calculated using an individual's weight and height. BMI provides a numerical value that categorizes individuals into different weight status categories, such as underweight, normal weight, overweight, or obese.
Insulin Sensitivity | Baseline assessment and at the final assessment at the end of the study (16 weeks)
  Blood draw test to obtain the homeostatic model assessment (HOMA-IR), an indirect method to quantify insulin resistance and pancreatic β-cell function. HOMA-IR is a mathematical model used to estimate insulin resistance based on fasting glucose and insulin levels. Higher values indicate higher insulin resistance therefore an improvement would be a lower value.
Sleep | Baseline assessment and at the final assessment at the end of the study (16 weeks)
  The 8-item PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep-Related Impairment questionnaire to measure alertness, sleepiness, tiredness, and functional impairments associated with sleep problems during waking hours.
  It assesses sleep disturbance over the past seven days. PROMIS instruments are scored using item-level calibrations on a 5 point likert scale from not at all to very much.
  Higher T-scores indicate greater sleep disturbance.
Body Composition: Waist circumference | Baseline assessment and at the final assessment at the end of the study (16 weeks)
  Waist circumference measures the circumference of the waist at a specific point, typically at the level of the natural waist or the midpoint between the lower rib and the iliac crest. Lower values indicate better health.
Respiratory Parameters | Baseline assessment, during the 6 minute walk test and at the final assessment at the end of the study (16 weeks)
  Spirometry to assess the forced expiratory volume in 1 second (FEV1). FEV1 is crucial for evaluating lung function and respiratory and global health. A higher value indicates better respiratory function
Respiratory Parameters | Baseline assessment, during the 6 minute walk test and at the final assessment at the end of the study (16 weeks)
  Spirometry to assess the forced expiratory flow (FEF). FEF is crucial for evaluating lung function and respiratory and global health. A higher value indicates better respiratory function.
Respiratory Parameters | Baseline assessment, during the 6 minute walk test and at the final assessment at the end of the study (16 weeks)
  Spirometry to assess the peak expiratory flow (PEF). PEF is crucial for evaluating lung function and respiratory and global health. A higher value
Respiratory Parameters | Baseline assessment, during the 6 minute walk test and at the final assessment at the end of the study (16 weeks)
  Spirometry to assess the maximal voluntary ventilation (MVV). MVV is crucial for evaluating lung function and respiratory and global health. A higher value would indicate better lung function.
Bowel and bladder management (BSS) | Baseline assessment and at the final assessment at the end of the study (16 weeks)
  The Bristol Stool Scale categorizes stool consistency into seven distinct types, ranging from hard lumps (Type 1) to watery diarrhea (Type 7), based on visual descriptions and illustrations. The BSS provides a standardized and objective method for individuals to describe their stool consistency, facilitating communication with healthcare providers.

CONTACTS AND LOCATIONS:
Overall Officials: Noel Keijsers, Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Hengstdal, Ubbergen, Netherlands

IPD SHARING:
Plan to Share IPD: No